CLINICAL TRIAL: NCT00121914
Title: Treatment of Hepatocellular Carcinoma: A Randomized Controlled Study With Long-Acting Somatostatin Plus Percutaneous Ethanol Instillation (PEI) Versus Long-Acting Somatostatin Alone
Brief Title: Treatment of Hepatocellular Carcinoma: Long-Acting Somatostatin Plus Percutaneous Ethanol Instillation (PEI) Versus Long-Acting Somatostatin Alone
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Medical University of Vienna (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCC-327-2000
Record Dates: First submitted 2005-07-15; First posted 2005-07-21 (Estimated); Last update posted 2005-10-18 (Estimated); Status verified 2005-07

CONDITIONS: Carcinoma, Hepatocellular
Keywords: Carcinoma, Hepatocellular,; percutaneous ethanol instillation; long-acting somatostatin
MeSH Terms: conditions — Carcinoma, Hepatocellular

INTERVENTIONS:
Procedure: percutaneous ethanol instillation (PEI)

SUMMARY:
Hepatocellular carcinoma (HCC) is a consequence of liver cirrhosis. In early tumour stages, tumour resection or liver transplantation are therapeutic options; later tumour stages may be treated with locally ablative treatments such as percutaneous ethanol instillation (PEI), transarterial chemoembolization (TACE) or radio-frequency thermoablation. This randomized study investigates the effect of PEI on survival of patients with HCC. All patients will receive hormonal treatment (long-acting somatostatin intramuscularly [i.m.]) and will be randomized for treatment with PEI or no additional treatment.

DETAILED DESCRIPTION:
This is a randomized two-arm parallel group study.

* Study group: PEI + long-acting somatostatin
* Control group: long-acting somatostatin alone

Aims of the study:

* Does treatment with PEI+ long-acting somatostatin prolong survival as compared to treatment with long-acting somatostatin alone?
* Can time to tumour progression be extended in patients treated with PEI + long-acting somatostatin as compared to treatment with long-acting somatostatin alone?

ELIGIBILITY:
Inclusion Criteria:

* Histologically-proven hepatocellular carcinoma
* Treatable with percutaneous ethanol instillation
* Inoperable tumour
* Age 18-85 years

Exclusion Criteria:

* Liver cirrhosis Child C
* Tumour diameter > 8 cm

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2000-10; Study Completion 2005-07

PRIMARY OUTCOMES:
survival time
time to tumour progression

SECONDARY OUTCOMES:
quality of life
causes of death

CONTACTS AND LOCATIONS:
Overall Officials: Christian Mueller, MD, Principal Investigator — Universitaetsklinik fuer Innere Medizin IV
Locations (1):
- Universitaetsklinik fuer Innere Medizin IV / Gastroenterologie und Hepatologie, Vienna, Vienna, Austria

REFERENCES:
- [Derived] Muller C, Schoniger-Hekele M, Schernthaner R, Renner B, Peck-Radosavljevic M, Brichta A, Wrba F, Posch M, Bauer P, Ferenci P, Gangl A. Percutaneous ethanol instillation therapy for hepatocellular carcinoma - a randomized controlled trial. Wien Klin Wochenschr. 2008;120(19-20):608-18. doi: 10.1007/s00508-008-1086-2. PMID 19083165